CLINICAL TRIAL: NCT06179082
Title: Efficacy of Polydioxanone Threads for Forehead Wrinkle Correction
Brief Title: Threads Insertion in Forehead Static Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Norhan Anees, Principal Investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: forehead wrinkles
Record Dates: First submitted 2023-12-19; First posted 2023-12-21 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Wrinkle

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): received Botox then threads
  Interventions: Combination Product: Botox then threads
- Group B (Active Comparator): received threads insertion only
  Interventions: Procedure: threads only

INTERVENTIONS:
Combination Product: Botox then threads — patients in which Botox injection then threads insertion were used
  Arms: Group A
Procedure: threads only — patients in which threads insertion only was used
  Arms: Group B

SUMMARY:
The main objective of this study is to analyze the efficacy and safety of PDO threads in correcting deep static wrinkles on the upper face.

DETAILED DESCRIPTION:
The upper face is a complex and dynamic part of the face, which conveys facial expression and emotion. As one age, youthful dynamic facial lines on the forehead and glabella change to static wrinkles, which remain on the face at rest. These permanent wrinkles can lead to the appearance of fatigue and negative facial expressions such as anger, which may influence psychological wellbeing, social confidence, and self-esteem.

The two major factors involved in the formation of static wrinkles in the upper face are repetitive muscle contraction and aging (loss of dermal collagen and matrix material leading to reduced dermal support). Compared with other facial muscles, the frontalis and corrugator muscles usually retain their muscle volume and even undergo hypertrophy to compensate for age-related ptosis and loss in visual acuity, which intensify the wrinkles.

Botulinum toxin and filler injections are currently the main treatment modalities in the management of facial wrinkles, especially for those on the upper third of the face. Conceptually, botulinum toxin addresses wrinkles by relaxing the muscles responsible for their creation (ie, the"dynamic" component), while soft tissue fillers provide necessary volume for the effacement of facial rhytids (ie, the "static" component). Although popular and widely accepted by the general population, some hesitate to receive toxin or filler injections due to the potential risk of unnatural facial expression, ptosis (associated with botulinum toxin), skin necrosis, and vision loss (from filler injection).

This has created a demand for a minimally invasive technique with reduced side effects, where threads may be considered. Although more commonly known as a mean for facial lifting, polydioxanone (PDO) suture materials have been applied to static wrinkles with promising outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult females and males between 30 and 65 years of age seeking treatment for static wrinkles on forehead.

Exclusion Criteria:

* • Patients who received filler injection within a period of 12 months before thread insertion and during the follow-up period.

  * Patients with a history of plastic surgery on the face.
  * Visible scars that may affect evaluation of a response and/or quality of photography and previous botulinum toxin treatment within the prior 12 months.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
improvement in wrinkles | 2 months after the procedure
  a Global Aesthetic Improvement Scale (GAIS) as follows: 1: no change; 2: improved; 3: much improved; 4: very much improved.
patient satisfaction | 2 months after the procedure
  using the following scale: excellent, very good, good, fair

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university hospitals, Zagazig, Egypt